CLINICAL TRIAL: NCT00002026
Title: Treatment and Suppression of Hairy Leukoplakia in ARC Patients With Oral Acyclovir (ACV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 033A; 179
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-05

CONDITIONS: Leukoplakia, Hairy; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Leukoplakia, Oral; Herpesvirus 4, Human; Acyclovir; AIDS-Related Complex
MeSH Terms: conditions — Leukoplakia, Hairy; HIV Infections; AIDS-Related Opportunistic Infections; Leukoplakia, Oral; Epstein-Barr Virus Infections; AIDS-Related Complex | interventions — Acyclovir

INTERVENTIONS:
Drug: Acyclovir

SUMMARY:
To evaluate the efficacy of oral acyclovir for the treatment and suppression of Epstein-Barr virus (EBV) related hairy leukoplakia (HL). To determine the long-term safety of acyclovir in the AIDS-related complex (ARC) patient with HL. To monitor the progression of HIV disease in the HL patient and compare to existing historical control data.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical antifungal therapy.

Patient must have:

* Newly diagnosed clinical and histological hairy leukoplakia.
* Positive HIV antibody by licensed ELISA or Western blot.

Exclusion Criteria

Co-existing Condition:

Patients with AIDS or a history of intolerance or allergy to acyclovir are excluded.

Concurrent Medication:

Excluded within 2 weeks of study entry:

* Systemic antifungal treatment.
* Excluded within 6 weeks of study entry:
* Immunomodulators.
* Systemic antiviral treatment.

Patients with AIDS or a history of intolerance or allergy to acyclovir are excluded.

Prior Medication:

Excluded within 2 weeks of study entry:

* Systemic antifungal.
* Excluded within 6 weeks of study entry:
* Immunomodulators.
* Systemic antiviral treatment.
* Excluded within 8 weeks of study entry:
* Zidovudine (AZT) or other antiretroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of Southern California / LA County USC Med Ctr, Los Angeles, California, United States

REFERENCES:
- [Background] Herbst JS, Morgan J, Raab-Traub N, Resnick L. Comparison of the efficacy of surgery and acyclovir therapy in oral hairy leukoplakia. J Am Acad Dermatol. 1989 Oct;21(4 Pt 1):753-6. doi: 10.1016/s0190-9622(89)70250-4. PMID 2808791